CLINICAL TRIAL: NCT03705156
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase III Clinical Trial Evaluating the Efficacy and Safety of ZL-2306 (Niraparib) for Maintenance Treatment in Patients With Platinum-sensitive Relapsed Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Cancer (Collectively Referred to as Ovarian Cancer)
Brief Title: Clinical Trial Evaluating the Efficacy and Safety of ZL-2306 (Niraparib) in Ovarian Cancer Patient
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL-2306-001
Record Dates: First submitted 2018-09-19; First posted 2018-10-15 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Platinum-sensitive Relapsed Ovarian Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZL-2306 (Experimental): The starting dose is 300 mg or 200 mg based on patient's body weight.
  Interventions: Drug: ZL-2306(nirapairb)
- Placebo (Placebo Comparator): The starting dose is the matched dose of placebo (3 capsules or 2 capsules).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ZL-2306(nirapairb) — The starting dose is 300 mg or 200 mg based on patient's body weight.
  Arms: ZL-2306
Drug: Placebos — The starting dose is the matched dose of placebo (3 capsules or 2 capsules).
  Arms: Placebo

SUMMARY:
This is a 2:1 randomized, double-blind, placebo-controlled, multi-center, phase III clinical study evaluating the efficacy and safety of ZL-2306 (niraparib) for maintenance treatment in patients with platinum-sensitive relapsed ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer (collectively referred to as relapsed ovarian cancer).The evaluation will be divided into two stages: Stage I will be conducted in all patients, and if the predetermined statistically significant difference is not reached, the trial will continue to extend to Stage II during which evaluation will be performed in gBRCA mutation-positive ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older female.
* High-grade serous or dominantly high-grade serous ovarian cancer
* The subject shall have received two lines of platinum-containing chemotherapy, complete response [CR] or partial response [PR] after first-line platinum-containing chemotherapy, and after received at least 4 cycles of platinum-containing (must be carboplatin or cisplatin or nedaplatin) in second-line platinum-containing chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Patients who have undergone ascites drainage with the last two cycles of the last chemotherapy regimen prior to enrollment.
* Symptomatic brain metastases or leptomeningeal metastases that have not been controlled.
* Patients who have been diagnosed previously or currently with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 265 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 35 months
  It is defined as the time from randomization to progressive disease or death due to various causes, whichever occurs first. Progressive disease will be determined by the Independent Central Imaging Review according to standard RECIST 1.1.

SECONDARY OUTCOMES:
Chemotherapy-free interval (CFI) | 35 months
  It refers to the time from the last platinum-containing treatment to the start of the next anti-cancer treatment (excluding maintenance treatment);
Time to first subsequent anti-cancer treatment (TFST) | 35 months
  It refers to the time from the date of randomization in the study to the date when the first subsequent anti-tumor treatment starts.
Overall survival (OS) | 35 months
  It refers to the time from the date of randomization to death for any cause.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Cancer center of Guangzhou medical university, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical university cancer hospital, Harbin, Heilongjiang
  - the first affiliated hospital of of Harbin medical university, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South Hospital, Changsha, Hunan
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The first Bethune Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shaanxi Cancer Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China second university hospital, Chengdu, Sichuan
  - Affiliate Cancer Hospital Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Woman's hospital School of medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Cancer hospital Chinese academy of medical science, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai
  - Tianjin Tumour Hospital, Tianjin

REFERENCES:
- [Derived] Wu X, Zhu J, Yin R, Yang J, Liu J, Wang J, Wu L, Liu Z, Gao Y, Wang D, Lou G, Yang H, Zhou Q, Kong B, Huang Y, Chen L, Li G, An R, Wang K, Zhang Y, Yan X, Lu X, Lu W, Hao M, Wang L, Cui H, Chen Q, Abulizi G, Huang X, Tian X, Wen H, Huang Z, Dong J, Zhang C, Hou J, Mirza MR. Niraparib maintenance therapy using an individualised starting dose in patients with platinum-sensitive recurrent ovarian cancer (NORA): final overall survival analysis of a phase 3 randomised, placebo-controlled trial. EClinicalMedicine. 2024 May 7;72:102629. doi: 10.1016/j.eclinm.2024.102629. eCollection 2024 Jun. PMID 38745967
- [Derived] Wu XH, Zhu JQ, Yin RT, Yang JX, Liu JH, Wang J, Wu LY, Liu ZL, Gao YN, Wang DB, Lou G, Yang HY, Zhou Q, Kong BH, Huang Y, Chen LP, Li GL, An RF, Wang K, Zhang Y, Yan XJ, Lu X, Lu WG, Hao M, Wang L, Cui H, Chen QH, Abulizi G, Huang XH, Tian XF, Wen H, Zhang C, Hou JM, Mirza MR. Niraparib maintenance therapy in patients with platinum-sensitive recurrent ovarian cancer using an individualized starting dose (NORA): a randomized, double-blind, placebo-controlled phase III trial☆. Ann Oncol. 2021 Apr;32(4):512-521. doi: 10.1016/j.annonc.2020.12.018. Epub 2021 Jan 14. PMID 33453391